CLINICAL TRIAL: NCT05868967
Title: A Clinical Study to Investigate the Mass Balance and Biotransformation of [14C]DWP14012 in Healthy Chinese Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Collaborators: Shanghai Haini Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DW_DWP14012112
Record Dates: First submitted 2023-04-07; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Phase 1 Study, Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: A single-center, single-dose, open-label design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]DWP14012 (Experimental): Type: [14C]DWP14012 suspension containing 40 mg/80 μCi Dosage: orally take the suspension
  Interventions: Drug: [14C]DWP14012

INTERVENTIONS:
Drug: [14C]DWP14012 — Each subject will receive a single oral dose of [14C]DWP14012 suspension (containing approximately 40 mg/80 μCi [14C]DWP14012) under fasting conditions.

SUMMARY:
The purpose of this study is to investigate the Mass Balance and Biotransformation of [14C]DWP14012 in Healthy Chinese Male Subjects

DETAILED DESCRIPTION:
This study is a single-center, single-dose, non-randomized, open-label design with two parts. Each subject will receive a single oral dose of [14C]DWP14012 suspension (containing approximately 40 mg/80 μCi [14C]DWP14012) under the fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 18 to 45 years (including boundary values);
2. Body weight ≥ 50.0 kg and body mass index (BMI) between 19.0 and 26.0 kg/m2 (including boundary values);
3. Subjects must give informed consent to this study before the study and voluntarily sign a written informed consent form;
4. Have no plan for fertility/sperm donation during the study and within 1 year after completion of the study, and take strict contraceptive measures with their spouses (see Appendix 3 for details);
5. Have good hygiene habits, and are able to communicate well with the investigator and complete the study in accordance with the study regulations.

Exclusion Criteria:

1. Subjects with an allergic constitution, including those with a history of drug allergy or allergic reactions and are known to be allergic to this product or other P-CABs, PPIs or other drugs (e.g., aspirin and antibiotics); and those who are allergic to any food ingredients or have special requirements for diet and unable to take the unified diet;
2. Subjects with clinically significant abnormalities or medical history of hepatic, renal, gastrointestinal, neurological, respiratory, endocrine, hematological, oncological, cardiovascular, urological, or psychiatric disorders;
3. Subjects with abnormal and clinically significant results of vital signs, physical examination, laboratory tests (hematology, blood chemistry, urinalysis, coagulation function, thyroid functions (FT3, FT4, TSH), stool routine + occult blood), 12-lead electrocardiogram, abdominal B-ultrasound (hepatobiliary, pancreas, spleen and kidney) as judged by the investigator;
4. Subjects who are positive for any one of the hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, and HIV antigen/antibody combination test (primary screening);
5. Subjects with any medical condition that, in the opinion of the investigator, may increase the risk during the subject's participation in this study (especially a history of esophageal or gastrointestinal ulcers), may interfere with drug absorption, distribution, metabolism or excretion, or may impair protocol compliance;
6. Subjects with frequent alcohol consumption within 6 months prior to screening, i.e., more than 14 units of alcohol per week (1 unit = 285 mL of beer or 25 mL of spirits containing 40% alcohol or 100 mL of wine); or alcoholics; or those with a positive alcohol breath test at screening and baseline admission;
7. Subjects who have smoked more than 5 cigarettes per day or habitually used nicotine-containing products within 3 months before screening and are unable to withdraw during the study;
8. Subjects who have used soft drugs (e.g., cannabis) within 3 months before screening or hard drugs (e.g., cocaine, amphetamines, phencyclidine, etc.) within 1 year before screening; or have a history of drug abuse; or have a positive urine drug test at screening and baseline admission;
9. Subjects who have taken any investigational product or participated in any clinical trial of drugs within 3 months prior to screening;
10. Subjects who have participated in blood donation within 3 months prior to screening with a total blood donation of ≥ 400 mL or total blood loss of ≥ 400 mL, or who have participated in blood donation within one month prior to screening with a total blood donation of ≥ 200 mL or total blood loss of ≥ 200 mL; or who have received blood transfusion; or who plan to donate blood within 1 month after the end of this study;
11. Subjects who have used any medication that alters liver enzyme activity within 4 weeks prior to dosing (see Appendix 1 for details);
12. Subjects who have used any prescription or over-the-counter drugs, any vitamin products, health care drugs or Chinese herbal medicines within 14 days prior to dosing;
13. Subjects who have habitual consumption of grapefruit juice or excessive amounts of tea, coffee and/or caffeine-containing beverages, and are unable to withdraw during the study;
14. Subjects with a history of fear of needles and hemophobia, difficulty in blood collection or intolerance to venipuncture blood collection; radiopharmaceutical labeling studies;
15. Subjects whose work requires long-term exposure to radioactive conditions; or who have significant radioactive exposure (≥ 2 chest/ abdominal CTs, or ≥ 3 other types of X-rays) within 1 year prior to screening; or who have participated in radiopharmaceutical labeling studies;
16. Subjects with other factors that are not suitable for participation in this study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Tmax | Up to 168hours(approx) from administration
  Time to peak Concentration
Cmax | Up to 168hours(approx) from administration
  Maximum Concentration
AUC0-t | Up to 168hours(approx) from administration
  Area under the plasma concentraion-time curve
AUC0-∞ | Up to 168hours(approx) from administration
  Area under the curve from time 0 extrapolated to infinite time
t1/2 | Up to 168hours(approx) from administration
  Elimination Phase Half-life
MRT | Up to 168hours(approx) from administration
  Mean Residence Time
CL/F | Up to 168hours(approx) from administration
  apparent oral clearnace
Vd/F | Up to 168hours(approx) from administration
  apparent oral volume of distribution
Ratio of total radioactivity in whole blood/plasma | Up to 168hours(approx) from administration
  Total measured radioactivity content of urine and fecal samples collected at each sampling interval
Cumulative recovery of total radioactive substances | Up to 168hours(approx) from administration
  Measurement of cumulative recovery ratio in urine or/and feces to meet the criteria for termination

SECONDARY OUTCOMES:
To observe the safety of [14C]DWP14012 | Up to study completion, approximately up to 2000 hours
  Adverse events, serious adverse events etc.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Hou, Principal Investigator — Beijing GoBroad Boren Hospital; Wel Tan, Principal Investigator — Beijing GoBroad Boren Hospital
Locations (1):
- Beijing GoBroad Boren Hospital, Beijing, China